CLINICAL TRIAL: NCT02123758
Title: A Drug-Drug Interaction, Safety and Efficacy Study With JNJ-56021927 (ARN-509) and Abiraterone Acetate in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of JNJ-56021927 (ARN-509) and Abiraterone Acetate in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR104358; 56021927PCR1010 (Other: Janssen Research & Development, LLC); 2014-001426-14 (EudraCT Number)
Record Dates: First submitted 2014-04-21; First posted 2014-04-28 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms; Metastatic Castration-Resistant Prostate Cancer
Keywords: Prostatic Neoplasms; Metastatic Castration-Resistant Prostate Cancer (mCRPC); Prostate cancer; Abiraterone Acetate (ZYTIGA); Prednisone; JNJ-56021927
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive abiraterone acetate (AA) along with prednisone on Day 1, Treatment Cycle 1 up to Day 7, Treatment Cycle 1; followed by combined intake of abiraterone acetate + prednisone (AAP) + JNJ-56021927 from Day 8, Treatment Cycle 1 up to the end of treatment (EoT) visit (ie, up to approximately 18 months). On Day 8, Treatment Cycle 2 participants will receive JNJ-56021927, 1 hour after intake of AA and prednisone. Breakfast will be offered approximately 30 minutes after intake of JNJ-56021927. Treatment cycles will be of 28 days.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: JNJ-56021927
- Cohort 2 (Experimental): Participants will receive abiraterone acetate (AA) along with prednisone on Day 1, Treatment Cycle 1 up to Day 7, Treatment Cycle 1; followed by combined intake of AAP + JNJ-56021927 from Day 8, Treatment Cycle 1 up to the end of treatment (EoT) visit (ie, up to approximately 18 months). On Days 7 and 36, participants will receive AA and prednisone together. On Day 8, Treatment Cycle 2 participants will receive JNJ-56021927, 1 hour after intake of AAP. Treatment cycles will be of 28 days.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: JNJ-56021927

INTERVENTIONS:
Drug: Abiraterone Acetate — Administered orally (by mouth) once daily in morning at a dose of 1000 mg for up to the end of treatment (EoT) visit (ie, for up to approximately 18 months).
  Other Names: ZYTIGA
Drug: Prednisone — Administered orally twice a day at a dose of 5mg for up to the end of treatment (EoT) visit (ie, for up to approximately 18 months).
Drug: JNJ-56021927 — Administered orally once daily in morning at a dose of 240 mg starting on Day 8, Treatment Cycle 1 for up to the end of treatment (EoT) visit (ie, for up to approximately 18 months).

SUMMARY:
The purpose of this study is to investigate potential drug-drug interaction (DDI) between JNJ-56021927 and abiraterone acetate and between JNJ-56021927 and prednisone, determine safety of the combination and evaluate in a descriptive manner the efficacy in these participants. It will also, potentially provide dosing recommendations for abiraterone acetate in future studies when combined with JNJ-56021927.

DETAILED DESCRIPTION:
This is a multicenter, open-label (participants will know the identity of study drug received) study in participants with Metastatic Castration-Resistant Prostate Cancer (mCRPC). The study is a single sequence design (ie, all participants will take abiraterone acetate + prednisone [AAP] once daily on Days 1-7 of Treatment Cycle 1 and then proceed with combined daily intake of AAP+JNJ-56021927 from Treatment Cycle 1, Day 8 through to the end of treatment [ie, for up to an expected duration of approximately 18 months] and will be conducted as two cohorts (group of participant's). The study will consist of a 28-day screening phase to determine eligibility, an open-label treatment phase consisting of 28-day treatment cycles, and a 30-day follow-up phase for collection of adverse events (AE) after last dose of study drug. Participants will have blood samples collected during the study to evaluate pharmacokinetics, safety, and antitumor activity (PSA). Participant safety will also be monitored by the collection of adverse events. Imaging assessments for disease evaluation will be planned at discretion of the Investigator. Once all participants have completed study treatment up to Cycle 3 Day 1, a data cutoff is planned to evaluate the short term safety profile of the combination and to complete the PK analysis up to the cutoff date. All participants will continue on study (ie, to receive treatment) until disease progression, withdrawal of consent, lost to follow-up, or the occurrence of unacceptable toxicity. The end of the study is defined when all participants have completed treatment. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Documentation of metastatic disease
* Prostate cancer progression
* Surgically or medically castrated, with testosterone levels of less than (<) 50 nanogram per deciliter (ng/dL)
* Adequate bone marrow and organ function

Exclusion Criteria:

* Known brain metastases
* Pathological finding consistent with small cell carcinoma of the prostate
* Administration of an investigational agent within 4 weeks of Treatment Cycle 1, Day 1
* Chemotherapy, or immunotherapy for the treatment of prostate cancer within 4 weeks of Treatment Cycle 1, Day 1
* Therapies that must be discontinued or substituted prior to Treatment Cycle 1, Day 1 include the following: Medications known to lower the seizure threshold; Herbal and non-herbal products that may decrease prostate specific antigen (PSA) levels (that is, saw palmetto, pomegranates or pomegranate juice); Medications known to induce drug metabolizing enzymes such as dexamethasone, rifampicin, carbamazepine, phenytoin, phenobarbital, St. John's wort, etc.; and, potent inhibitors of CYP3A4 or CYP2C8

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time Zero to Time 24 Hours (AUC [0-24]) of abiraterone | Day 7 (Treatment Cycle 1) and on Day 36 (Treatment Cycle 2)
  The AUC (0-24) is area under the plasma concentration-time curve from time zero to time 24 hours.
Maximum plasma concentration (Cmax) of abiraterone, prednisone and its metabolite prednisolone | Day 7 (Treatment Cycle 1) and on Day 36 (Treatment Cycle 2)
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Time 12 Hours (AUC [0-12]) of prednisone and its metabolite prednisolone | Day 7 (Treatment Cycle 1) and on Day 36 (Treatment Cycle 2)
  The AUC (0-12) is area under the plasma concentration-time curve from time zero to time 12 hours.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Curve (AUC [0- 24h]) of JNJ-56021927 and its metabolite JNJ-56142060 | Day 36 (Treatment Cycle 2), on Day 57 (Treatment Cycle 3)
  The AUC (0-24) is area under the plasma concentration-time curve from time zero to time 24 hours.
Maximum plasma concentration (Cmax) of JNJ-56021927 and its metabolite JNJ-56142060 | Day 36 (Treatment Cycle 2), on Day 57 (Treatment Cycle 3)
  The Cmax is the maximum observed plasma concentration.
Change in prostate specific antigen (PSA) | Up to the end of the treatment phase (approximately 18 months)
  Prostate-specific antigen (PSA) is a protein produced by cells of the prostate gland.
Maximal decline in prostate specific antigen (PSA) | Up to the end of the treatment phase (approximately 18 months)
  Prostate-specific antigen (PSA) is a protein produced by cells of the prostate gland.

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc. Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (7):
- United States (3):
  - Los Angeles, California
  - San Francisco, California
  - Houston, Texas
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec
- Rotterdam, Netherlands
- Sutton, United Kingdom